CLINICAL TRIAL: NCT03580005
Title: A Phase 4, Double-blind, Randomized, Parallel Group, Placebo-controlled Study Of The Efficacy And Safety Of Quillichew (Methylphenidate Hydrochloride (Hcl)) Extended Release Chewable Tablets (Erct) In 4-5 Year Old Children With Attention Deficit Hyperactivity Disorder (Adhd)
Brief Title: A 6-week Study to Evaluate the Safety and Efficacy of Quillichew ERCT in 4-5 Year Old Children With ADHD.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was cancelled prior to the enrollment of any participants.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7491019
Record Dates: First submitted 2018-05-16; First posted 2018-07-09 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Quillichew ERCT (Active Comparator): Quillichew ERCT
  Interventions: Drug: methylphenidate HCl ERCT
- Placebo to match Quillichew ERCT (Placebo Comparator): Placebo to match Quillichew ERCT
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: methylphenidate HCl ERCT — methylphenidate HCl ERCT
  Arms: Quillichew ERCT
Drug: Placebo — Placebo to Match Quillichew ERCT
  Arms: Placebo to match Quillichew ERCT

SUMMARY:
A 6-week double-blind study to evaluate the safety and efficacy of Quillichew extended release chewable tablets in 4-5 year old children with attention deficit hyperactivity disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female child 4-5 years of age at baseline.
2. Signed and dated informed consent document.
3. Meets DSM-V criteria for ADHD based on the K-SADS-PL.
4. ADHD RS-IV Preschool Home Version score at Screening and Baseline >/= 90th percentile for gender and age in >/=1 of the following: hyperactive-impulsive subscale, inattentive subscale, or total score.
5. Peabody Picture Vocabulary Test 4 (PPVT4)Standard Score >/=70.
6. Child Global Assessment Scale (CGAS) score </= 55.

Exclusion Criteria:

1. Treated with atomoxetine within 30 days prior to the Baseline.
2. Received any investigational products or devices within 30 days prior to the Baseline visit.
3. History of stimulant nonresponse, intolerability or hypersensitivity to any dose of Quillichew ERCT or other stimulant.
4. An intelligence quotient (IQ) <70.
5. History of acute or chronic medical or psychiatric condition or cardiac or laboratory abnormality.
6. Less than 5th percentile for height or weight at Screening.
7. History of recent clinically significant self-harming behaviors.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-10-31 (Estimated); Primary Completion 2021-10-12 (Estimated); Study Completion 2021-10-12 (Estimated)

PRIMARY OUTCOMES:
Safety-incidence of treatment emergent adverse events | 6 months
  incidence of treatment emergent adverse events
Attention Deficit Hyperactivity Rating Scale - IV (ADHD RS-IV) Preschool-Home Version | 6 weeks
  Change from Baseline to end of double-blind treatment in the total score of the Attention Deficit Hyperactivity Rating Scale - IV (ADHD RS-IV) Preschool-Home Version

SECONDARY OUTCOMES:
incidence of adverse events | 6 weeks
  incidence of adverse events
Clinical Global Impression of Improvement (CGI-I) Scale Score | weeks 1-6
  CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Clinician responded to a question: "Compared to your subject's condition at the beginning of treatment, how much has your subject changed?". Improvement was compared to baseline and was defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Intellectual Performance of Children Using Child Behavior Checklist 4-18 Years (CBCL 4-18) | Weeks 1-6
  CBCL was standardized for children ages 4 to 18 years and measured child internalizing and externalizing behaviors and total problems. The 4-18 years' checklist contains 140 questions and responses were recorded on a Likert scale: 0 = Not True, 1 = Somewhat or Sometimes True, 2 = Very True or Often True. The range of possible values was 0-280 (0=good to 280=worst).
Children's Global Assessment Scale (CGAS) | Week 6
  CGAS: clinician-rated global assessment item for children based on symptoms and social functioning in home, school, and community settings. Scores on this single item range from 1 (most impaired) to 100 (healthiest); higher levels indicate greater health, with descriptive anchors for every 10-point interval. Scores above 70 on this scale are considered within the "normal" range; lower score indicates need for increased supervision.
Mean Clinical Global Impression - Severity (CGI-S) score | Weeks 1-6
  CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491019&StudyName=A+6-month+Open-label+Extension+Study+Of+Protocol+B7491017
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491019&StudyName=A+Phase+4%2C+6-month+Open+Label+Extension+Study+To+Evaluate+The+Safety%2C+Tolerability+And+Efficacy+Of+Quillichew+Extended+Release+Chewable+Tablets+%28methylphenidate+Hcl+Extended+Release+Chewable+Tablets+%5Berct%5D%29+In+Children+With+Attention+Deficit+Hyperactivity+Disorder+%28adhd%29+Who+Participated+In+Study+B7491017+Or+Study+B7491020.
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491019&StudyName=A+Phase+4%2C+6-month+Open-label+Extension+Study+To+Evaluate+The+Safety%2C+Tolerability+And+Efficacy+Of+Quillichew+%28methylphenidate+Hydrochloride+%28hcl%29%29+Extended+Release+Chewable+Tablets+%28erct%29+In+Children+With+Attention+Deficit+Hyperactivity+Disorder+%28adhd%29+Who+Participated+In+Study+B7491017+Or+Study+B7491020.
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491017&StudyName=A+Multi-center%2C+Double-blind%2C+Randomized%2C+Placebo-controlled%2C+Parallel+Group+Study+Evaluating+The+Safety+And+Efficacy+Of+Quillivant+Xr+In+The+Treatment+Of+Pre-school+Aged+Children+With+Adhd
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491017&StudyName=A+Phase+4%2C+Double-blind%2C+Randomized%2C+Parallel+Group%2C+Placebo-controlled+Study+Of+The+Efficacy+And+Safety+Of+Quillichew+Extended+Release+Chewable+Tablets+%28methylphenidate+Hcl+Extended+Release+Chewable+Tablets+%28erct%29%29++In+4-5+Year+Old+Children+With+Attention+Deficit+Hyperactivity+Disorder+%28adhd%29.
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491017&StudyName=A+Phase+4%2C+Double-blind%2C+Randomized%2C+Parallel+Group%2C+Placebo-controlled+Study+Of+The+Efficacy+And+Safety+Of+Quillichew+%28methylphenidate+Hydrochloride+%28hcl%29%29+Extended+Release+Chewable+Tablets+%28erct%29+In+4-5+Year+Old+Children+With+Attention+Deficit+Hyperactivity+Disorder+%28adhd%29